CLINICAL TRIAL: NCT05092555
Title: Clinical Presentations and Outcomes of Patients With Covid-19 Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ghada Mohamed Bahy, Chest resident, Sohag University
Other Study IDs: Soh-Med-21-10-24
Record Dates: First submitted 2021-10-22; First posted 2021-10-25 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: COVID-19 Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Nasopharyngeal swap for Reverse transcription polymerase chain reaction — Nasopharyngeal swap and Blood sample is taken for doing previous tests and CT chest is done for all patients
  Other Names: CT chest d-dimer C-reactive protein serum ferritin

SUMMARY:
This study aims at determining clinical presentations and outcomes of patients with covid-19 pneumonia and also follow up of patients for up to 6 months to detect possibility of post covid fibrosis

DETAILED DESCRIPTION:
According to the World Health Organization (WHO), the emergence of viral diseases represents a serious public health risk. In the past two decades, several epidemics caused by viruses such as the severe acute respiratory syndrome coronavirus (SARS-CoV) from 2002 to 2003, and H1N1 influenza in 2009, and the Middle East respiratory syndrome coronavirus (MERS-CoV) in 2012 have been described which have had a significant impact on global health. Since being declared a global pandemic by the WHO, SARS-CoV-2, the virus responsible for COVID-19 has spread to 223 countries with more than 178 million confirmed cases, and more than 3.8 million deaths reported worldwide. The U.S. experienced the highest number of SARS-CoV-2 infections and COVID-19 related deaths followed by Brazil and India.

In fact, COVID-19 was the third leading cause of death in the U.S. in 2020 after heart disease and cancer, with approximately 375,000 death reported . As of 22 June 2021, the Alpha(B.1.1.7) variant has spread to 170 countries, the Beta (B.1.351) variant has been reported in 119 countries, the Gamma (P.1) variant has been detected in 71 countries and the Delta variant(B.1.617.2) has spread to 85 countries around the world based on the weekly epidemiological update by the WHO . The WHO's current estimate of the global case fatality rate for COVID-19 is 2.2%. However, the case fatality rate is affected by factors that include age, underlying preexisting conditions, and severity of illness and significantly varies between countries.

The common clinical features of COVID-19 pneumonia in adults include fever, dry cough, sore throat, headache, fatigue, myalgia and breathlessness . The disease manifestations in the infected patients range from mild pneumonia (81%) to moderate pneumonia (hypoxia requiring hospitalization, 14%), and critical illness (leading to invasive mechanical ventilation, multiorgan dysfunction and possibly death, 5%). The risk of death depends on age, underlying comorbidities and severity of the disease, increasing up to 49% in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Patients with covid-19 pneumonia confirmed by:

Reverse transcription polymerase chain reaction Or pattern of covid-19 in computed tomography (CT) scan ( ground-glass opacity indicative of pneumonia on CT, opinion on consolidation, etc) with laboratory investigations

Exclusion Criteria:

1. Patients not confirmed to be covid-19 with PCR or radiologically.
2. Patients who are diagnosed as bacterial pneumonia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with covid-19 pneumonia
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Post covid fibrosis | Six month
  Possibility of occurrence of post covid fibrosis by follow up of patients for up to 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy A Mohammadeen, Ass.prof, Study Director — Sohag University; Mona T Hussen, Ass.prof, Study Chair — Sohag University